CLINICAL TRIAL: NCT00671905
Title: Circumferential vs Ganglionated Plexi Ablation in Patients With Paroxysmal Atrial Fibrillation: A Randomized Study
Brief Title: Circumferential Versus Ganglionated Plexi Ablation for Atrial Fibrillation (AF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiovascular Research Society, Greece (Other)
Responsible Party: Principal Investigator, Dr D Katritsis, Dr Demosthenes Katritsis, MD, PhD(Lon), FRCP, FESC, FACC, Cardiovascular Research Society, Greece
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1. 25/4/08
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; PV isolation; ablation; ganglionic plexi; parasympathetic denervation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Circumferential PV isolation
  Interventions: Procedure: PV isolation
- 2 (Active Comparator): HF stimulation-guided and anatomic ablation of the main right and left atrial GP.
  Interventions: Procedure: GP ablation
- 3 (Active Comparator): HF stimulation-guided and anatomic ablation of the main right and left atrial GP followed by circumferential PV isolation
  Interventions: Procedure: GP ablation; Procedure: PV isolation

INTERVENTIONS:
Procedure: GP ablation — HF stimulation-guided and anatomic ablation of the main right and left atrial GP
  Arms: 2; 3
Procedure: PV isolation — Circumferential PV isolation
  Arms: 1; 3

SUMMARY:
The investigators have recently shown that anatomic ganglionated plexi (GP) ablation is inferior to circumferential pulmonary vein (PV) ablation for the treatment of paroxysmal AF. In this study, however, 26% of patients subjected to GP ablation alone without circumferential lesions were free of AF-recurrence up to one year after the ablation procedure. The investigators hypothesized that a combination of circumferential ablation with high-frequency-stimulation-identified GP ablation is superior to conventional circumferential ablation for the prevention of recurrences of paroxysmal atrial fibrillation (AF). The investigators are, therefore, conducting a randomized study comparing conventional circumferential ablation to a combination of circumferential ablation plus specific right and left atrial GP ablation in patients with drug-refractory paroxysmal AF.

DETAILED DESCRIPTION:
Introduction:

In clinical studies, epicardial or endocardial partial ganglionated plexi (GP) ablation may prevent AF,1-4 and parasympathetic denervation has been proposed as a potential mechanism of circumferential or antral pulmonary vein (PV) ablation for the treatment of atrial fibrillation.5,6 However, there have also been reports of a temporary only 7 or even proarrhythmic effect of this approach by means of increased vulnerability of vagally-mediated AF,8,9 or ablation-related macro-reentrant left atrial tachycardias.10 Thus, the potential contribution of GP modification to clinical success of circumferential or antral pulmonary vein ablation that unavoidably affects adjacent GP is not known. Few publications exist on isolated GP ablation with variable results in terms of eliminating paroxysmal or persistent AF.11-13 We have recently shown that anatomically-oriented regional ablation at the areas of GP is superior to selective GP ablation, following identification of GP by high-frequency stimulation, conferring success rates comparable to these of pulmonary vein (PV) isolation procedures.13 We hypothesized that GP ablation guided by both HF stimulation and anatomical orientation is superior to PV isolation in patients with paroxysmal AF. We also aimed at comparing these two approaches with a combination of GP ablation and PV isolation. We are, therefore, conducting a randomized study comparing the three techniques in patients with drug-refractory paroxysmal AF.

Methods:

Patients with symptomatic, paroxysmal AF were randomized to three groups:

Group 1. Patients are subjected to conventional PV isolation through circumferential ablation 1-2 cm from the PV ostium.

Group 2. Patients are subjected to specific, HF stimulation-guided and anatomic ablation of the main right and left atrial GP.

Group 3. Patients are subjected to specific, HF stimulation-guided and anatomic ablation of the main right and left atrial GP followed by PV isolation.

Group 1. PV isolation. Circumferential ablation around the antra of the PV with the aid of electroanatomical mapping (Carto, Biosence-Webster) at a distance of approximately 1-2 cm from the ostia of the left and right PVs (46°C, 35W, 17 mL/min, Stockert, Biosense Webster), aimed at a voltage reduction by > 80% or a peak to peak bipolar electrogram <0.1 mV. End-point of both approaches is verification of PV isolation with demonstration of entry and exit block. The area encircled by circumferential ablation will be calculated using the software provided by the CARTO system.

Group 2. GP ablation. The anatomic areas of GP are identified in the right and left atrium. Anatomic locations of GP were considered around the PV: anterior right (ARGP), inferior right (IRGP), left superior (LSGP), and left inferior GP (LIGP). In addition the following GP were considered: The GP at the crux of the left atrium which is probably near or in continuation with the IRGP (2-3 cm below the lower edge of RIPV), expanding both toward the mitral annulus and inferior aspect of the LA posterior wall (cruxGP). This GP was also approached from the crux of the RA, behind the tendon of Tadaro/Eustachian ridge and the coronary sinus ostium. The GP at the septal-posterior aspect of the junction of the RA with the SVC (this GP may actually correspond to the 3rd fat pad located at the junction of SVC-RA-right PA-aorta).14-18 Following anatomic orientation, precise determination of the location of parasympathetic GP is accomplished by high-frequency stimulation.19 Patients are deeply sedated with diamorphine and diazepam without intubation, and high-frequency stimulation is delivered with a Grass stimulator at 1,200 bpm (20 Hz) with a pulse width of 10 ms at 20 V. A predominant parasympathetic response is defined as induction of AV block (> 2 sec) and hypotension or prolongation of the R-R interval by >50% during AF, following a 5 seconds application of high-frequency stimulation.19 Before applying high-frequency stimulation to inferior GP, extra care is taken to ensure that the catheter tip is not on the annulus to avoid induction of ventricular fibrillation. Verification of catheter position is accomplished by examination of recorded electrograms and anatomic location on both lateral views on CARTO. The sequence of GP ablation is: LS GP, LI GP, ARGP GP, IRGP, right anterior GP and the crux GP situated in the RA. After each ablation lesion (46°C, 35W for 60 seconds, 17 mL/min), parasympathetic response is reassessed by high-frequency stimulation. End-point for radiofrequency delivery is abolition of parasympathetic response. Following specific GP ablation, anatomical ablation is performed as previously described, in a way that the designated anatomic areas of GP are ablated.

Group 3. GP ablation and PV isolation. Following specific and anatomic GP ablation as previously described, PV isolation is accomplished either by circumferential or antral ablation.

At the end of the ablation procedure in both groups, AF or atrial flutter induction is attempted by isoproterenol infusion and high left atrial pacing. Induction of atrial fibrillation is registered but does not necessitate additional ablation. Induction of right, isthmus-dependent atrial flutter is dealt with cavotricuspid isthmus ablation. Left atrial flutters will be studied by means of entrainment from the mitral isthmus and the adjacent posterior wall. Since a considerable percentage of these arrhythmias disappear with time,20 they will be ablated only if sustained (> 3 minutes) and associated with 1:1 ventricular response.

Follow-up. Patients will be prospectively assessed for recurrence of AF or other atrial arrhythmia. As part of our routine AF ablation protocol, all patients are receiving beta blockers, whereas all patients are kept on amiodarone and warfarin for 3 months post-ablation. Patients will be subjected to monthly clinical assessment and ambulatory electrocardiographic monitoring for 2 years. All patients are instructed to maintain personal records with descriptions of every episode of symptomatic palpitations and, in case of persistent arrhythmia episodes, to obtain trans-telephonic or electrocardiographic documentation of the underlying rhythm. Patients will be encouraged to use trans-telephonic monitoring even when their symptoms are not typical for recurrent AF. A successful outcome over the follow-up period is defined as the lack of electrocardiographically recorded AF, and no AF or other atrial arrhythmia on Holter, and subjective symptomatic improvement after a 3-month blanking period.

Heart rate variability will be measured at 6, 12, 18 and 24 months after ablation.

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal AF
* age < 75 years
* left atrial size < 5 cm

Exclusion Criteria:

* malignancies
* LVEF < 35%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Freedom of AF or other atrial arrhythmia | 2 years

SECONDARY OUTCOMES:
Quality of life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: D Katritsis, MD, Study Director — Cardiovascular Research Society; E Pokushalov, MD, Principal Investigator — State Research Institute of Circulation Pathology, Novosibirsk, Russia
Locations (2):
- Athens Euroclinic, Athens, Greece
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- [Background] Scanavacca M, Pisani CF, Hachul D, Lara S, Hardy C, Darrieux F, Trombetta I, Negrao CE, Sosa E. Selective atrial vagal denervation guided by evoked vagal reflex to treat patients with paroxysmal atrial fibrillation. Circulation. 2006 Aug 29;114(9):876-85. doi: 10.1161/CIRCULATIONAHA.106.633560. Epub 2006 Aug 21. PMID 16923757
- [Background] Schauerte P, Scherlag BJ, Pitha J, Scherlag MA, Reynolds D, Lazzara R, Jackman WM. Catheter ablation of cardiac autonomic nerves for prevention of vagal atrial fibrillation. Circulation. 2000 Nov 28;102(22):2774-80. doi: 10.1161/01.cir.102.22.2774. PMID 11094046
- [Background] Lemola K, Chartier D, Yeh YH, Dubuc M, Cartier R, Armour A, Ting M, Sakabe M, Shiroshita-Takeshita A, Comtois P, Nattel S. Pulmonary vein region ablation in experimental vagal atrial fibrillation: role of pulmonary veins versus autonomic ganglia. Circulation. 2008 Jan 29;117(4):470-7. doi: 10.1161/CIRCULATIONAHA.107.737023. Epub 2008 Jan 14. PMID 18195170
- [Background] McClelland JH, Duke D, Reddy R. Preliminary results of a limited thoracotomy: new approach to treat atrial fibrillation. J Cardiovasc Electrophysiol. 2007 Dec;18(12):1289-95. doi: 10.1111/j.1540-8167.2007.00977.x. Epub 2007 Oct 5. PMID 17919294
- [Background] Nakagawa H, Jackman WM, Scherlag BJ, Lazzara R. Pulmonary vein isolation during atrial fibrillation: insight into the mechanism of pulmonary vein firing. J Cardiovasc Electrophysiol. 2003 Mar;14(3):261-2. doi: 10.1046/j.1540-8167.2003.03002.x. No abstract available. PMID 12716107
- [Background] Pappone C, Santinelli V, Manguso F, Vicedomini G, Gugliotta F, Augello G, Mazzone P, Tortoriello V, Landoni G, Zangrillo A, Lang C, Tomita T, Mesas C, Mastella E, Alfieri O. Pulmonary vein denervation enhances long-term benefit after circumferential ablation for paroxysmal atrial fibrillation. Circulation. 2004 Jan 27;109(3):327-34. doi: 10.1161/01.CIR.0000112641.16340.C7. Epub 2004 Jan 5. PMID 14707026
- [Background] Oh S, Zhang Y, Bibevski S, Marrouche NF, Natale A, Mazgalev TN. Vagal denervation and atrial fibrillation inducibility: epicardial fat pad ablation does not have long-term effects. Heart Rhythm. 2006 Jun;3(6):701-8. doi: 10.1016/j.hrthm.2006.02.020. Epub 2006 Mar 6. PMID 16731474
- [Background] Hirose M, Leatmanoratn Z, Laurita KR, Carlson MD. Partial vagal denervation increases vulnerability to vagally induced atrial fibrillation. J Cardiovasc Electrophysiol. 2002 Dec;13(12):1272-9. doi: 10.1046/j.1540-8167.2002.01272.x. PMID 12521345
- [Background] Cummings JE, Gill I, Akhrass R, Dery M, Biblo LA, Quan KJ. Preservation of the anterior fat pad paradoxically decreases the incidence of postoperative atrial fibrillation in humans. J Am Coll Cardiol. 2004 Mar 17;43(6):994-1000. doi: 10.1016/j.jacc.2003.07.055. PMID 15028356
- [Background] Pokushalov E, Turov A, Shugayev P, Artyomenko S, Romanov A, Shirokova N. Catheter ablation of left atrial ganglionated plexi for atrial fibrillation. Asian Cardiovasc Thorac Ann. 2008 Jun;16(3):194-201. doi: 10.1177/021849230801600304. PMID 18515667
- [Background] Katritsis D, Giazitzoglou E, Sougiannis D, Goumas N, Paxinos G, Camm AJ. Anatomic approach for ganglionic plexi ablation in patients with paroxysmal atrial fibrillation. Am J Cardiol. 2008 Aug 1;102(3):330-4. doi: 10.1016/j.amjcard.2008.03.062. Epub 2008 May 22. PMID 18638596
- [Derived] Katritsis DG, Pokushalov E, Romanov A, Giazitzoglou E, Siontis GC, Po SS, Camm AJ, Ioannidis JP. Autonomic denervation added to pulmonary vein isolation for paroxysmal atrial fibrillation: a randomized clinical trial. J Am Coll Cardiol. 2013 Dec 17;62(24):2318-25. doi: 10.1016/j.jacc.2013.06.053. Epub 2013 Aug 21. PMID 23973694
- [Derived] Katritsis DG, Giazitzoglou E, Zografos T, Pokushalov E, Po SS, Camm AJ. Rapid pulmonary vein isolation combined with autonomic ganglia modification: a randomized study. Heart Rhythm. 2011 May;8(5):672-8. doi: 10.1016/j.hrthm.2010.12.047. Epub 2010 Dec 31. PMID 21199686